CLINICAL TRIAL: NCT06644729
Title: From Rotator Cuff Repair to Reverse Shoulder Arthroplasty - Clinical and Radiological Results
Status: Recruiting | Type: Observational
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: Sykehuset Telemark (Other Government); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Kjersti Kaul Jenssen, Principal Investigator, Lovisenberg Diakonale Hospital
Other Study IDs: CARS3
Record Dates: First submitted 2024-09-10; First posted 2024-10-16 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Tear Arthropathy; Rotator Cuff Injuries
Keywords: PROM; Rotator Cuff Repair; Rotator Cuff Tear; Cuff Arthropathy
MeSH Terms: conditions — Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 10 years after surgery: Cohort of 733 participants will be invited to a 10 year follow up and will be evaluated with patient reported outcome measurements and x-ray.
  Interventions: Procedure: Arthroscopic Rotator Cuff Repair

INTERVENTIONS:
Procedure: Arthroscopic Rotator Cuff Repair — Arthroscopic Rotator Cuff Repair

SUMMARY:
In the planned study the investigators will invite 733 participants 10 years after arthroscopic rotator cuff repair to a follow up examination.

Shoulder pain is a common problem in the Norwegian population. Rotator cuff tear is a major cause of shoulder pain with a reported prevalence of up to 51% in patients 60-80 years of age. Arthroscopic rotator cuff repair is performed in an increasing proportion of these patients. Good results in shoulder function has been reported, although there is a lack in published good quality studies and long term follow up of these patients. There is also a lack of evidence regarding the association between radiologically-verified re-tear and clinical outcome.

In this project, the investigators address these critical gaps in knowledge and aim to investigate the factors influencing the clinical outcome after rotator cuff surgery and re-tear in a large prospective cohort study. The investigators will investigate how many participants suffering from poor outcome and develop cuff arthropathy in need of reverse shoulder arthroplasty after 10 years.

DETAILED DESCRIPTION:
10 years after surgery: A cohort study of 733 participants with rotator cuff tear operated arthroscopically at Lovisenberg Diaconal Hospital during 2010-2014. The investigators will ask the participants included at the time of surgery to participate in a ten-year follow-up. The investigators will ask them to submit validated patient reported outcome measurements (PROMs): Western Ontario Rotator Cuff Index, EQ-5D-5L, Subjective Shoulder Value. The investigators will also evaluate the radiological result and signs of cuff arthropathy on x-ray according to Hamada-Fukuda and Seebauer classification.

The main objective is to quantify the relative importance of preoperative and perioperative prognostic factors on functional outcomes ten years after rotator cuff repair. The secondary objective is to identify and quantify patients who need shoulder replacement surgery ten years after rotator cuff surgery as a measure of failure.

ELIGIBILITY:
Inclusion Criteria:

* Operated at Lovisenberg Diaconal Hospital in the time period 2010-2014 with an arthroscopic rotator cuff repair
* Included in the rotator cuff registry at Lovisenberg Diaconal Hospital
* Able to read and write Norwegian

Exclusion Criteria:

* Lack of competence to consent
* Not able to submit patient reported outcome measurements in any way and not able to undergo x-ray
* Patient is unwilling to participate

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is participants with a rotator cuff repair treated with arthroscopic rotator cuff repair 2010-2014 at Lovisenberg Diaconal Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 733 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index, Norwegian Version | 10 Years after surgery
  Scale 0-2100. The maximum score is 2100 (higher score means worse outcome). Zero (0) represents no symptoms at all.

SECONDARY OUTCOMES:
Eurocol questionnaire EQ-5D-5L Norwegian version | 10 Years after surgery
  Standardized generic questionnaire measuring health in five dimensions. 5 health dimensions described above includes 5 response categories of no problem, slight problems, moderate problems, severe problems, and extreme problems. The 5 responses give a health state or profile represented by a 5-digit number (for example, 12231) corresponding to response categories reported by patients for successive dimensions
Subjective Shoulder Value | 10 Years after surgery
  A patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%.
Rotator cuff survival | 10 Years after surgery
  Survival of rotator cuff repair in terms of number of reverse shoulder arthroplasties performed in the study group
Cuff arthropathy | 10 years after surgery
  Developement of cuff arthropathy on x-ray by Hamada-Fukuda and Seebauer classification. X-ray will be conducted in one Y-view (scapular view), three anterioposterior view (with arm in neutral, 30 degrees of internal rotation and 60 degrees of external rotation).

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Kaul Jenssen, MD, PhD, Principal Investigator — Lovisenberg Diaconal Hospital
Locations (1):
- Lovisenberg Diacolan Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT06644729/Prot_SAP_000.pdf